CLINICAL TRIAL: NCT04947969
Title: Clinical Effect of Laser Acupuncture on Improving Cancer-related Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Wu Chung Hung, Chinese medicine department, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REC110-09
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cancer-related Fatigue
Keywords: Laser acupuncture

STUDY DESIGN:
Intervention Model Description: Randomized controlled, double blind, cross-over study.
Who Masked: Participant, Outcomes Assessor
Masking Description: After random assignment to 2 groups, patients in the RS and SR groups will receive real and shame laser acupuncture (single blinding), six consecutive times every day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rear laser acupuncture group (Experimental): Patients in the Real laser acupuncture group will receive real laser pen irradiation.
  Interventions: Device: laser acupuncture
- Shame laser acupuncture group (Sham Comparator): Patients in the Shame laser acupuncture group will receive shame laser pen irradiation.
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — This study will use German-made low-level laser pen (Al-Ga-As diode laser, 810nm, NIR, Physiolaser Olympic Basic, RJ laser). The parameters are power of 100mW, frequency of Bahr, apply on acupoint. Well will irradiate each point for 2 J. Each patient will receive this treatment six times for one week.

SUMMARY:
The aim of this study is to examine the clinical effect of laser acupuncture on improving cancer-related fatigue

DETAILED DESCRIPTION:
This study adopted a randomized controlled design, 2-arm trial cross-over study. All eligible patients included in the study agreed to participated and signed the informed consent from and the study procedures were approved by the ethical committee of Taichung Tzu Chi general hospital (REC110-09). Patients were recruited from the hematology oncology department of Taichung Tzu Chi general hospital. After random assignment to 2 groups, patients in the RS and SR groups will receive real and shame laser acupuncture. Before laser acupuncture, one week later, we will evaluate the patient-reported cancer-related fatigue index and other co-morbid symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 to 85 years old
* Patients who signed the informed consent form
* Patients who have been given a diagnosis of cancer
* Able to communicate verbally and completely fill the questionnaires

Exclusion Criteria:

* Patients who have given a diagnosis of cognitive impairment are unable to completely the questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue evaluation | 30 minutes
  ICD-10 Fatigue Criteria Brief Fatigue inventory-Taiwan Form
Cancer-related fatigue Assessment | 15 minutes
  Brief Fatigue Inventory-Taiwanese (BFI-T)

SECONDARY OUTCOMES:
Quality of Life Assessments | 15 minutes
  Functional Assessment of Cancer Therapy-general (FACT-G7)
Symptoms distress Assessments | 20 minutes
  Taiwanese Version of the M.D. Anderson symptom Inventory (MDASI-T)